CLINICAL TRIAL: NCT04605393
Title: Does Cannabidiol Attenuate the Acute Effects of ∆9-tetrahydrocannabinol Intoxication in Individuals Diagnosed With Schizophrenia? A Double-blind, Randomised, Placebo-controlled Experimental Study
Acronym: INTEGRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Edward Chesney, Psychiatrist/Clinical Research Fellow/Study Co-ordinator, King's College London
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRAS: 278595
Record Dates: First submitted 2020-10-05; First posted 2020-10-28 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia; Cannabis Use
MeSH Terms: conditions — Schizophrenia | interventions — Cannabidiol; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo/THC (Experimental): Oral placebo followed by inhalation of cannabis containing THC.
  Interventions: Drug: Placebo; Drug: Delta-9-THC
- CBD/THC (Experimental): Oral CBD 1000mg followed by inhalation of cannabis containing THC.
  Interventions: Drug: Cannabidiol; Drug: Delta-9-THC

INTERVENTIONS:
Drug: Cannabidiol — CBD
  Arms: CBD/THC
Drug: Placebo — Placebo
  Arms: Placebo/THC
Drug: Delta-9-THC — THC

SUMMARY:
This study will recruit schizophrenia patients who use cannabis recreationally. Each participant will attend the laboratory on three occasions: an initial visit to check that they are safe to join the study and two days of testing.

Participants will be administered, in a randomized order, a pre-treatment with either CBD (1000mg) orally or a matching placebo. On both experiments, participants will then inhale cannabis containing THC. The THC administration will follow a standardised inhalation procedure using a medical-grade vaporizer device.

Participants will complete a series of tasks measuring cognition, psychosis, anxiety and other subjective experiences.

The study will be carried out at the NIHR-Wellcome Trust Clinical Research Facility at King's College Hospital.

ELIGIBILITY:
Inclusion criteria:

* Age 18-65 years.
* Clinical diagnosis of schizophrenia (i.e. documented as such in the patient's clinical records and satisfying ICD-10 criteria for F20)
* Clinically stable for at least three months (since discharge from hospital, home treatment team, or prior clinical deterioration, and with agreement from the patient's responsible clinician)
* Regular (at least weekly) cannabis use for the past 3 months or more
* Evidence from either clinicians or from the patient that cannabis use exacerbates their symptoms or increases their risk of relapse
* Treatment with regular doses of antipsychotic medication for at least 1 month, confirmed by a blood test at the baseline visit, and with the participant agreeing to be maintained at a stable dose over the course of the experiment
* The participant agrees to abstain from cannabis use for at least 24hours prior to study visits
* The participant is willing to have an intravenous cannula inserted to collect blood samples on experimental visits
* Sufficiently fluent English
* Providing written informed consent

Exclusion criteria:

* Extreme cannabis use: participant is estimate to be using over 1gram of cannabis/day
* Dependence on alcohol or illicit substances other than cannabis as defined by ICD-10
* Pregnancy (current or planned) or breastfeeding
* Physical health disorder or another mental health disorder that the study psychiatrist judges may influence the patient's ability to tolerate the procedure, or that may alter the results of the study.
* Taken part in any drug study within the last 3 months or taking part in another study over the course of the trial
* Drug sensitivity/allergy to cannabis or Lorazepam
* Unlikely to be able to complete the study sessions for any reason, as judged by the study psychiatrist

Additional criteria which must be met on experimental visits:

* Negative alcohol breath test
* Negative urine drug screen (apart from cannabis and prescribed medication)
* Negative urine pregnancy test
* Stable mental state as judged by the study psychiatrist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test | Baseline visit; 20 mins post-THC
  Delayed verbal recall
Positive and Negative Syndrome Scale | pre-CBD/placebo administration, and from immediately after THC inhalation until the end of study visit (i.e. 2-3 hours post-THC)
  Positive Subscale

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | pre-CBD/placebo administration, pre-THC and 20mins post-THC
  State Scale
Digit span | Baseline; 25 mins post-THC
  Forward & Reverse
Hopkins Verbal Learning Test | Baseline; 20 mins post-THC
  Immediate verbal recall
Positive and Negative Syndrome Scale | pre-CBD/placebo administration, and from immediately after THC inhalation until the end of study visit (i.e. 2-3 hours post-THC)
  Negative Subscale
Visual analogue scales | pre-CBD/placebo, 90mins post CBD, pre-THC, and +10mins, +45mins, +90mins post-THC inhalation, and at the end of study visit (i.e. 2-3 hours post-THC)
  * Feel drug effect
  * Like drug effect
  * Want more drug
  * Thinking clearly
  * Tired
  * Excited
  * Want to talk
  * Anxious
  * Relaxed
  * Happy
  * Irritable
  * Suspicious
  * Hearing voices
  * Dry mouth
  * Hungry
Psychotomimetic states inventory | pre-CBD/placebo administration, and at the end of study visit (i.e. 2-3 hours post-THC)
State Social Paranoia Scale | pre-CBD/placebo administration, and at the end of study visit (i.e. 2-3 hours post-THC)
Study drug preference | End of Experiment 2
  At the end of the final experimental visit (i.e. 2-3 hours post-THC), participants will be asked to order the two experimental visits according to which drug combination they found most pleasurable.
Advice Taking Task | Baseline visit; 30 mins post-THC
White Noise Task | Baseline visit; 50 mins post-THC
Plasma delta-9-tetrahydrocannabinol (THC) concentration | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC
Plasma cannabidiol (CBD) concentration | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC
Plasma THC-COOH concentraion | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC
Plasma 11-COOH-THC concentration | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC
Plasma 11-OH-THC concentration | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC
Plasma 6-OH-CBD concentration | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC
Plasma anandamide concentration | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC
Plasma 2-arachidonoylglycerol concentration. | pre-CBD/placebo, 90mins post CBD, and 0mins, 5mins, 15mins, +90mins post-THC

CONTACTS AND LOCATIONS:
Overall Officials: Gill Dale, Study Chair — slam-ioppn.research@kcl.ac.uk
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chesney E, Oliver D, Sarma A, Lamper AD, Slimani I, Lloyd M, Dickens AM, Welds M, Krakstrom M, Gasparini-Andre I, Oresic M, Lawn W, Babayeva N, Freeman TP, Englund A, Strang J, McGuire P. Does cannabidiol reduce the adverse effects of cannabis in schizophrenia? A randomised, double-blind, cross-over trial. Neuropsychopharmacology. 2025 Nov;50(12):1759-1767. doi: 10.1038/s41386-025-02175-3. Epub 2025 Jul 24. PMID 40702165

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT04605393/Prot_SAP_002.pdf